CLINICAL TRIAL: NCT01817816
Title: Early Injection of Botulinum Toxin on Motor Function and Gait Pattern in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Ta-Sen Wei,MD, Director, Physical Medical and Rehabilitation, Principal Investigator, Clinical Professor, Changhua Christian Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CCH-061203
Record Dates: First submitted 2013-03-21; First posted 2013-03-25 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Stroke; Spasticity
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Botox_A (Experimental): receiving Botulinum Toxin Type-A (Botox-A, Allergan) at both affected lower extremity (aLE) and upper extremity (aUE)
  Interventions: Procedure: Botox_A
- placebo_A (Placebo Comparator): receiving placebo injection at both aLE & aUE ; receiving Botox-A at both aLE & aUE at 6-month.
  Interventions: Procedure: Botox_A
- Botox_B (Experimental): receiving Botox-A injection at aLE and placebo injection (sterile normal saline) at aUE.
  Interventions: Procedure: Botox_B
- placebo_B (Placebo Comparator): receiving placebo injection at both aLE & aUE ; receiving Botox-A only at aLE at 6-month.
  Interventions: Procedure: Botox_B

INTERVENTIONS:
Procedure: Botox_A
  Arms: Botox_A; placebo_A
Procedure: Botox_B
  Arms: Botox_B; placebo_B

SUMMARY:
Spasticity, muscle weakness, abnormal gait pattern are co-morbidities commonly seen in stroke patients. They cause disabled condition of patients in activities of daily life and functional performance, and also accidental falls and subsequent fractures.

This study is to evaluate and compare the effects of different phase injection of Botulinum Toxin Type-A at affected limbs on muscle rheological changes, muscle activity, muscle tone, functional performance, gait pattern and energy consumption in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* first-ever stroke, with spasticity within 3-months (MAS=2~3)
* independent walking 10 meters (with assistive devices)

Exclusion Criteria:

* recurrent stroke, cognition impaired
* lower limb fracture
* received anti-spasticity injection in the past

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-01; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in the muscle tone in upper and lower extremity | 4 weeks after injection
  use modified Ashworth Scale to access elbow, wrist, ankle joint muscle tone 0: normal
  1. slight hypertonus, at the end-range 1+: mild hypertonus, catch when limb is moved (<1/2)
  2. moderate hypertonus,, limbs moves easily (>1/2)
  3. passive movement difficult
  4. rigid

SECONDARY OUTCOMES:
Change in the gait pattern as walking | 4 weeks after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian Hospital, Dawan, Changhua, Taiwan